CLINICAL TRIAL: NCT04248075
Title: Effect of Sedatives on Perioperative Electroencephalogram in Elderly Patients Undergoing Spinal Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 20200120
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Effect of Sedatives
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Patients who do not want to be sedated during spinal anesthesia are included. Electroencephalogram is performed before, during, and 1 day after surgery.
  Interventions: Device: Electroencephalogram
- Dexmedetomidine: Patients who want to be sedated during spinal anesthesia are included. Electroencephalogram is performed before, during, and 1 day after surgery.
  After the induction of spinal anestheisa, dexmedetomidine is administered for sedation during surgery.
  Interventions: Device: Electroencephalogram
- Propofol: Patients who want to be sedated during spinal anesthesia are included. Electroencephalogram is performed before, during, and 1 day after surgery.
  After the induction of spinal anestheisa, propofol is administered for sedation during surgery.
  Interventions: Device: Electroencephalogram
- Midazolam: Patients who want to be sedated during spinal anesthesia are included. Electroencephalogram is performed before, during, and 1 day after surgery.
  After the induction of spinal anestheisa, midazolam is administered for sedation during surgery.
  Interventions: Device: Electroencephalogram

INTERVENTIONS:
Device: Electroencephalogram — Electroencephalogram is performed before, during, and 1 day after surgery in elderly patients undergoing spinal anesthesia.

SUMMARY:
In the present study, we observe perioperative findings of electroencephalogram in sedated and non-sedated elderly patients undergoing total knee arthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
In the present study, we observe perioperative findings of electroencephalogram in sedated and non-sedated elderly patients undergoing total knee arthroplasty under spinal anesthesia. Electroencephalogram is performed before, during, and 1 day after surgery.

After the induction of anesthesia, sedation is performed according to the patient's request. If a patient want to be sedated during surgery, one of the three sedatives (dexmedetomidine, propofol, and midazolam) is administered.

ELIGIBILITY:
Inclusion Criteria:

* Eldery patients scheduled for spinal anesthesia

Exclusion Criteria:

* MMSE ≤ 23
* Hemodynamic unstability
* Liver disease
* Renal disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients scheduled to undergo total knee arthroplasty under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-02-20 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
EEG frequency bands (alpha, beta, theta, delta, and gamma waves) during spinal anesthesia | 30 min after the induction of spinal anesthesia
  EEG frequency bands are observed during spinal anesthesia under sedated or unsedated states.

SECONDARY OUTCOMES:
EEG frequency bands (alpha, beta, theta, delta, and gamma waves) 1 day after surgery | 1 day after surgery
  EEG frequency bands are observed after surgery and compared with the preoperative findings.
Incidence of delirium | For 7 days after surgery.
  Delirium is assessed after surgery.